CLINICAL TRIAL: NCT01538940
Title: Randomized Controlled Trial to Compare the Immunogenicity of Intramuscular Versus Intradermal Trivalent Inactivated Split Virion Influenza Vaccine in HIV-infected Men Who Have Sex With Men in Bangkok, Thailand
Brief Title: Immunogenicity of Influenza Vaccines in HIV-infected Persons in Thailand
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDC-NCIRD-6181; 1U01GH000152 (NIH)
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Influenza
Keywords: Influenza; Vaccine; Thailand
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- HIV+, CD4<200, ID vaccine (Active Comparator): Humoral and cell-mediated immune responses among HIV-infected individuals with CD4 cell counts less than 200 per microliter will be compared to immune responses in HIV-infected individuals with CD4 cell counts of 200 per microliter or greater.
  Interventions: Biological: Intradermal vaccine
- HIV+, CD4<200, IM vaccine (Active Comparator): Humoral and cell-mediated immune responses among HIV-infected individuals with CD4 cell counts less than 200 per microliter will be compared to immune responses in HIV-infected individuals with CD4 cell counts of 200 per microliter or greater.
  Interventions: Biological: Intramuscular vaccine
- HIV+, CD4>=200, ID vaccine (Active Comparator): Humoral and cell-mediated immune responses among HIV-infected individuals with CD4 cell counts less than 200 per microliter will be compared to immune responses in HIV-infected individuals with CD4 cell counts of 200 per microliter or greater.
  Interventions: Biological: Intradermal vaccine
- HIV+, CD4 >=200, IM vaccine (Active Comparator): Humoral and cell-mediated immune responses among HIV-infected individuals with CD4 cell counts less than 200 per microliter will be compared to immune responses in HIV-infected individuals with CD4 cell counts of 200 per microliter or greater.
  Interventions: Biological: Intramuscular vaccine
- HIV-, ID vaccine (Other): A small HIV-uninfected MSM control group will be enrolled (with persons randomized into either an intramuscular or intradermal TIV arm) to serve as a comparator group for the cell-mediated immunity studies.
  Interventions: Biological: Intradermal vaccine
- HIV-, IM vaccine (Other): A small HIV-uninfected MSM control group will be enrolled (with persons randomized into either an intramuscular or intradermal TIV arm) to serve as a comparator group for the cell-mediated immunity studies.
  Interventions: Biological: Intramuscular vaccine

INTERVENTIONS:
Biological: Intradermal vaccine — 15ug
  Arms: HIV+, CD4<200, ID vaccine; HIV+, CD4>=200, ID vaccine; HIV-, ID vaccine
Biological: Intramuscular vaccine — 15ug
  Arms: HIV+, CD4 >=200, IM vaccine; HIV+, CD4<200, IM vaccine; HIV-, IM vaccine

SUMMARY:
This study will assess the efficacy of a new intradermal formulation of the trivalent inactivated influenza vaccine compared to the standard intramuscular vaccine in HIV-infected men who have sex with men in Bangkok, Thailand. Relative efficacy of the two different formulations of influenza vaccine will be assessed by comparing immunologic responses to vaccine between the two study arms.

DETAILED DESCRIPTION:
This study will assess the efficacy of a new intradermal formulation of the trivalent inactivated influenza vaccine (TIV) compared to standard intramuscular TIV in HIV-infected men who have sex with men (MSM) in Bangkok, Thailand. Eligible participants will be randomized to receive standard full-dose intramuscular vaccine versus full-dose intradermal vaccine. Full dose (15 micrograms) intradermal TIV will be licensed for use in adult's ≥ 60 years of age in Thailand in mid-2011. In this study, intradermal TIV will be used off-label as the 15 microgram dose will be administered to individuals < 60 years of age. Efficacy of the two different formulations of influenza vaccine will be assessed by comparing immunologic responses to vaccine between the two HIV-infected study arms. Both humoral (influenza antibody) and cell-mediated (influenza- specific CD4 and CD8 T cell) immune responses will be evaluated. Humoral and cell-mediated immune responses among HIV-infected individuals with CD4 cell counts less than 200 per microliter will also be compared to immune responses in HIV-infected individuals with CD4 cell counts of 200 per microliter or greater. A small HIV-uninfected MSM control group will also be enrolled (with persons randomized into either an intramuscular or intradermal TIV arm) to serve as a comparator group for the cell-mediated immunity studies.

ELIGIBILITY:
Inclusion Criteria:

* Thai men by nationality who have sex with men
* HIV-infected or HIV-uninfected men
* At least 18 years of age
* Willing and able to provide written informed consent
* Availability and commitment for 12 months of study follow-up (3 study visits)

Exclusion Criteria:

* Men with severe allergies to chicken eggs (they will specifically be asked about severe egg allergies during the screening visit; appendix C1)
* Men > 60 years of age
* Men who have had a severe reaction to influenza vaccine in the past
* Men with a history of Guillain-Barré Syndrome
* Men who received influenza vaccine within 12 months prior to enrollment
* Men who are on steroid therapy or other immunosuppressant medications
* Men who received any vaccine in the 4 weeks prior to the first study visit or who plan to receive a vaccine (other than influenza vaccine provided through the study protocol) in the 4 weeks following the first study visit
* Men who received an experimental agent (vaccine, drug, biologic, device, blood product, medication) within 1 month prior to enrollment in this study, or expect to receive an experimental agent during the 12 month study period
* Men who have any condition, in the opinion of the investigator, that would place them at an unacceptable risk of injury or render them unable to meet requirements of the protocol. (e.g., severe reaction to another vaccine, blood clotting disorder, inflammatory skin condition).
* Foreign (non-Thai) nationality

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 415 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2013-09-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Antibody titers | 30 days
  Frequency of 4-fold or greater increase in serum hemagglutination inhibition antibody titers against each viral strain in the vaccine

SECONDARY OUTCOMES:
Antibody titers | 6 months
  Frequency of 4-fold or greater increase in serum hemagglutination inhibition antibody titers against each viral strain in the vaccine
Antibody titers | 12 months
  Frequency of 4-fold or greater increase in serum hemagglutination inhibition antibody titers against each viral strain in the vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Charung Muangchana, MD, Principal Investigator — Ministry of Health, Thailand; Prasert Thongcharoen, MD, Principal Investigator — Influenza Foundation of Thailand
Locations (1):
- Silom Community Clinic, Bangkok, Thailand

REFERENCES:
- [Derived] Amoah S, Mishina M, Praphasiri P, Cao W, Kim JH, Liepkalns JS, Guo Z, Carney PJ, Chang JC, Fernandez S, Garg S, Beacham L, Holtz TH, Curlin ME, Dawood F, Olsen SJ, Gangappa S, Stevens J, Sambhara S. Standard-Dose Intradermal Influenza Vaccine Elicits Cellular Immune Responses Similar to Those of Intramuscular Vaccine in Men With and Those Without HIV Infection. J Infect Dis. 2019 Jul 31;220(5):743-751. doi: 10.1093/infdis/jiz205. PMID 31045222
- [Derived] Garg S, Thongcharoen P, Praphasiri P, Chitwarakorn A, Sathirapanya P, Fernandez S, Rungrojcharoenkit K, Chonwattana W, Mock PA, Sukwicha W, Katz JM, Widdowson MA, Curlin ME, Gibbons RV, Holtz TH, Dawood FS, Olsen SJ. Randomized Controlled Trial to Compare Immunogenicity of Standard-Dose Intramuscular Versus Intradermal Trivalent Inactivated Influenza Vaccine in HIV-Infected Men Who Have Sex With Men in Bangkok, Thailand. Clin Infect Dis. 2016 Feb 1;62(3):383-391. doi: 10.1093/cid/civ884. Epub 2015 Oct 20. PMID 26486702
- See also: Website for clinic where the study is being conducted. — http://www.silomclinic.in.th/